CLINICAL TRIAL: NCT04915495
Title: The Use of the LuViva Advanced Cervical Scan to Identify Women at High-Risk for Cervical Neoplasia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Guided Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CC-03-01-2020
Record Dates: First submitted 2021-05-28; First posted 2021-06-07 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cervical Dysplasia
Keywords: Cervical cancer, dysplasia, detection
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Singe-arm Study (Experimental): Experimental device being evaluated for sensitivity and specificity.
  Interventions: Diagnostic Test: LuViva Advanced Cervical Scan

INTERVENTIONS:
Diagnostic Test: LuViva Advanced Cervical Scan — Multimodal hyperspectral device

SUMMARY:
This study is designed to demonstrate that a multimodal hyperspectral device (LuViva) is able to segregate women with abnormal screening tests into Low and High risk groups for the purpose of determining whether they require enhanced colposcopy and additional biopsies in order to increase detection of CIN2+ cervical disease.

DETAILED DESCRIPTION:
This study is a matched pair design, single-arm study with the following two treatments: current standard of care (SOC) and the LuViva study device. After undergoing the LuViva test, all study subjects will first undergo the SOC (i.e., nominal) colposcopy, with the colposcopist noting on the case report form (CRF), locations of lesions with colposcopy impression of CIN1+. Then the colposcopist will employ enhanced colposcopy measures that include the use on Lugol's solution and green/blue filters. The colposcopist will note on the CRF any additional lesions that became evident as a result of these enhanced measures, regardless of colposcopic impression. Biopsies of these lesions will be taken. Biopsies identified using SOC practices will be placed in vials labeled "SOC Samples". Biopsies identified using enhanced practices will be placed in vials labeled "Additional Samples". The colposcopist will then take a biopsy from any quadrant at the squamocolumnar junction (SCJ) in which a lesion was not observed. These biopsies will be placed in the vial labeled "Additional Samples". Once all colposcopy procedures are completed, biopsies of lesions collected, and biopsies of any non-lesion identified quadrants collected, an ECC, if indicated, will be collected. If an ECC would have been taken per SOC practices, it will be placed in a vial labeled "SOC ECC". ECCs collected per enhanced procedures will be placed in a vial labeled "Additional ECC". The study is a matched pair design because all subjects are tested with the LuViva device, and all will undergo both the nominal (minimal) colposcopy and biopsy treatment pursuant to ASCCP Guidelines as well as enhanced colposcopy and biopsy. By analyzing all biopsy specimens from SOC procedures and enhanced procedures, it can be determined 1) Whether enhanced procedures can be justified when the LuViva test indicates High-risk by the increase in detection of CIN2+ and 2) That when LuViva indicates Low-risk, that enhanced procedures (in the absence of a LuViva High-risk result) are not the reason for increased detection of CIN2+. Subjects will be enrolled during their normally scheduled colposcopy visit and will be recruited from the pool of patients that are referred to colposcopy based on the ASCCP Guidelines published in April 2020. The total number of enrolled female subjects pooled across all clinical sites combined will not exceed 500 in order to target an evaluable cohort of approximately 400 women.

ELIGIBILITY:
Inclusion Criteria:

* Able to read or understand and give informed consent
* Referral Pap test within 120 days
* Scheduled for colposcopy based on the 2019 ASCCP Management Guidelines that fall within the 4% to 59% Immediate CIN3+ risk with the exception of women who lack a cervix or may be pregnant and are recommended to colposcopy.*

  * Notes: The rationale for defining the referral inclusion criteria as women scheduled for colposcopy is that this group has been identified with having a significant likelihood of being diagnosed with CIN2+ over the two year period after being referred to colposcopy because of an abnormal screening test or tests. For example, the ALTS results showed that women with ASC-US plus high-risk HPV, LSIL, ASC-H, AGC and HSIL all had a likelihood of CIN2+ of approximately 10% to 20% or greater in the cases of ASC-H and HSIL (5). More recently, it has been shown that this threshold also carries with it a 4% or greater likelihood of immediate CIN3+ (12).

Exclusion Criteria:

* Pregnancy
* Menstruating on the day of colposcopy and LuViva test
* Radiation therapy to her genitourinary system within 1 year
* Prior hysterectomy in which cervix was removed
* Congenital anatomical cervical variant (e.g., double cervix)
* Friable cervix at the time of the study (i.e., a cervix that bleeds easily upon minimal contact or trauma)
* Post-coital or other significant bleeding at the time of the exam
* Excessive cervical mucous or discharge that cannot be removed and is significant enough, in the opinion of the Investigator, to interfere with a Pap test or colposcopy, resulting from inflammation, bacterial infection or other sources
* History of any photosensitizing disease or other disease affected by Ultra-violet radiation, (e.g., pophyria, Lupus Erythematosus).
* Undergoing phototherapy
* Recent use of photosensitizing agents, such as fluoroquinolones or retinoids
* Under-screened populations - defined as those women who have not been screened within the past 5 years who also screen positive for any HPV genotype

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Diagnostic Device | up to 60 days after completion of enrollment
  LuViva's ability to correctly identify diseased tissue. LuViva result indicated High-risk and the pathology results indicate the presence of disease cervical tissue.

SECONDARY OUTCOMES:
Specificity of Diagnostic Device | up to 60 days after completion of enrollment
  LuViva's ability to correctly identify non diseased tissue. LuViva result indicated Low-risk and the pathology results did not indicate the presence of disease cervical tissue.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama Birmingham- Heersink School of Medicine, Birmingham, Alabama
  - Emory University- Winship Cancer Institute, Atlanta, Georgia
  - Great Lakes Bay Health Centers, Bay City, Michigan
  - Tidewater Clinical Research, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Sherman ME, Schiffman M, Cox JT; Atypical Squamous Cells of Undetermined Significance/Low-Grade Squamous Intraepithelial Lesion Triage Study Group. Effects of age and human papilloma viral load on colposcopy triage: data from the randomized Atypical Squamous Cells of Undetermined Significance/Low-Grade Squamous Intraepithelial Lesion Triage Study (ALTS). J Natl Cancer Inst. 2002 Jan 16;94(2):102-7. doi: 10.1093/jnci/94.2.102. PMID 11792748
- [Background] Wright TC Jr, Cox JT, Massad LS, Twiggs LB, Wilkinson EJ; ASCCP-Sponsored Consensus Conference. 2001 Consensus Guidelines for the management of women with cervical cytological abnormalities. JAMA. 2002 Apr 24;287(16):2120-9. doi: 10.1001/jama.287.16.2120. PMID 11966387
- [Background] ASCUS-LSIL Traige Study (ALTS) Group. Results of a randomized trial on the management of cytology interpretations of atypical squamous cells of undetermined significance. Am J Obstet Gynecol. 2003 Jun;188(6):1383-92. doi: 10.1067/mob.2003.457. PMID 12824967
- [Background] Massad LS, Collins YC. Strength of correlations between colposcopic impression and biopsy histology. Gynecol Oncol. 2003 Jun;89(3):424-8. doi: 10.1016/s0090-8258(03)00082-9. PMID 12798706
- [Background] Mitchell MF, Schottenfeld D, Tortolero-Luna G, Cantor SB, Richards-Kortum R. Colposcopy for the diagnosis of squamous intraepithelial lesions: a meta-analysis. Obstet Gynecol. 1998 Apr;91(4):626-31. doi: 10.1016/s0029-7844(98)00006-4. PMID 9540955
- [Background] Wentzensen N, Massad LS, Mayeaux EJ Jr, Khan MJ, Waxman AG, Einstein MH, Conageski C, Schiffman MH, Gold MA, Apgar BS, Chelmow D, Choma KK, Darragh TM, Gage JC, Garcia FAR, Guido RS, Jeronimo JA, Liu A, Mathews CA, Mitchell MM, Moscicki AB, Novetsky AP, Papasozomenos T, Perkins RB, Silver MI, Smith KM, Stier EA, Tedeschi CA, Werner CL, Huh WK. Evidence-Based Consensus Recommendations for Colposcopy Practice for Cervical Cancer Prevention in the United States. J Low Genit Tract Dis. 2017 Oct;21(4):216-222. doi: 10.1097/LGT.0000000000000322. PMID 28953109
- [Background] Twiggs LB, Chakhtoura NA, Ferris DG, Flowers LC, Winter ML, Sternfeld DR, Lashgari M, Burnett AF, Raab SS, Wilkinson EJ. Multimodal hyperspectroscopy as a triage test for cervical neoplasia: pivotal clinical trial results. Gynecol Oncol. 2013 Jul;130(1):147-51. doi: 10.1016/j.ygyno.2013.04.012. Epub 2013 Apr 13. PMID 23591399
- [Background] Huh WK, Papagiannakis E, Gold MA. Observed Colposcopy Practice in US Community-Based Clinics: The Retrospective Control Arm of the IMPROVE-COLPO Study. J Low Genit Tract Dis. 2019 Apr;23(2):110-115. doi: 10.1097/LGT.0000000000000454. PMID 30694884
- [Background] Perkins RB, Guido RS, Castle PE, Chelmow D, Einstein MH, Garcia F, Huh WK, Kim JJ, Moscicki AB, Nayar R, Saraiya M, Sawaya GF, Wentzensen N, Schiffman M; 2019 ASCCP Risk-Based Management Consensus Guidelines Committee. 2019 ASCCP Risk-Based Management Consensus Guidelines for Abnormal Cervical Cancer Screening Tests and Cancer Precursors. J Low Genit Tract Dis. 2020 Apr;24(2):102-131. doi: 10.1097/LGT.0000000000000525. No abstract available. PMID 32243307
- [Background] Cheung LC, Egemen D, Chen X, Katki HA, Demarco M, Wiser AL, Perkins RB, Guido RS, Wentzensen N, Schiffman M. 2019 ASCCP Risk-Based Management Consensus Guidelines: Methods for Risk Estimation, Recommended Management, and Validation. J Low Genit Tract Dis. 2020 Apr;24(2):90-101. doi: 10.1097/LGT.0000000000000528. PMID 32243306
- [Background] Waxman AG, Conageski C, Silver MI, Tedeschi C, Stier EA, Apgar B, Huh WK, Wentzensen N, Massad LS, Khan MJ, Mayeaux EJ Jr, Einstein MH, Schiffman MH, Guido RS. ASCCP Colposcopy Standards: How Do We Perform Colposcopy? Implications for Establishing Standards. J Low Genit Tract Dis. 2017 Oct;21(4):235-241. doi: 10.1097/LGT.0000000000000336. PMID 28953112
- [Background] Jeronimo J, Schiffman M. Colposcopy at a crossroads. Am J Obstet Gynecol. 2006 Aug;195(2):349-53. doi: 10.1016/j.ajog.2006.01.091. Epub 2006 May 3. PMID 16677597
- [Background] Gage JC, Hanson VW, Abbey K, Dippery S, Gardner S, Kubota J, Schiffman M, Solomon D, Jeronimo J; ASCUS LSIL Triage Study (ALTS) Group. Number of cervical biopsies and sensitivity of colposcopy. Obstet Gynecol. 2006 Aug;108(2):264-72. doi: 10.1097/01.AOG.0000220505.18525.85. PMID 16880294
- [Background] Nam K, Chung S, Kwak J, Cha S, Kim J, Jeon S, Bae D. Random biopsy after colposcopy-directed biopsy improves the diagnosis of cervical intraepithelial neoplasia grade 2 or worse. J Low Genit Tract Dis. 2010 Oct;14(4):346-51. doi: 10.1097/LGT.0b013e3181e9635b. PMID 20885163
- [Background] Pretorius RG, Belinson JL. Colposcopy. Minerva Ginecol. 2012 Apr;64(2):173-80. PMID 22481626
- [Background] Pretorius RG, Belinson JL, Azizi F, Peterson PC, Belinson S. Utility of random cervical biopsy and endocervical curettage in a low-risk population. J Low Genit Tract Dis. 2012 Oct;16(4):333-8. doi: 10.1097/LGT.0b013e3182480c18. PMID 22622343
- [Background] van der Marel J, van Baars R, Rodriguez A, Quint WG, van de Sandt MM, Berkhof J, Schiffman M, Torne A, Ordi J, Jenkins D, Verheijen RH, Helmerhorst TJ, Ter Harmsel B, Wentzensen N, Del Pino M. The increased detection of cervical intraepithelial neoplasia when using a second biopsy at colposcopy. Gynecol Oncol. 2014 Nov;135(2):201-7. doi: 10.1016/j.ygyno.2014.08.040. Epub 2014 Sep 7. PMID 25204846
- [Background] Wentzensen N, Walker JL, Gold MA, Smith KM, Zuna RE, Mathews C, Dunn ST, Zhang R, Moxley K, Bishop E, Tenney M, Nugent E, Graubard BI, Wacholder S, Schiffman M. Multiple biopsies and detection of cervical cancer precursors at colposcopy. J Clin Oncol. 2015 Jan 1;33(1):83-9. doi: 10.1200/JCO.2014.55.9948. Epub 2014 Nov 24. PMID 25422481
- [Background] Baasland I, Hagen B, Vogt C, Valla M, Romundstad PR. Colposcopy and additive diagnostic value of biopsies from colposcopy-negative areas to detect cervical dysplasia. Acta Obstet Gynecol Scand. 2016 Nov;95(11):1258-1263. doi: 10.1111/aogs.13009. PMID 27564523
- [Background] Hu SY, Zhang WH, Li SM, Li N, Huang MN, Pan QJ, Zhang X, Han Y, Zhao FH, Chen W, Qiao YL. Pooled analysis on the necessity of random 4-quadrant cervical biopsies and endocervical curettage in women with positive screening but negative colposcopy. Medicine (Baltimore). 2017 Apr;96(17):e6689. doi: 10.1097/MD.0000000000006689. PMID 28445270
- [Background] Stoler MH, Vichnin MD, Ferenczy A, Ferris DG, Perez G, Paavonen J, Joura EA, Djursing H, Sigurdsson K, Jefferson L, Alvarez F, Sings HL, Lu S, James MK, Saah A, Haupt RM; FUTURE I, II and III Investigators. The accuracy of colposcopic biopsy: analyses from the placebo arm of the Gardasil clinical trials. Int J Cancer. 2011 Mar 15;128(6):1354-62. doi: 10.1002/ijc.25470. PMID 20506504
- [Background] Sawaya GF, Kuppermann M. Identifying a "range of reasonable options" for cervical cancer screening. Obstet Gynecol. 2015 Feb;125(2):308-310. doi: 10.1097/AOG.0000000000000670. No abstract available. PMID 25569012